CLINICAL TRIAL: NCT01780038
Title: Smokers' Response to Nicotine Dependence Genotyping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0069-12-FB
Record Dates: First submitted 2013-01-25; First posted 2013-01-30 (Estimated); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Cigarette Smoking; Nicotine Dependence
Keywords: Cigarette Smoking; Nicotine Dependence; Smoking Abstinence; Health Literacy; Genetic Predisposition Testing; Heredity
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receipt of Genetic Results (Experimental): Receipt of Genetic Results indicates that participants have received the results of genotyping for RS1051730
  Interventions: Behavioral: Receipt of Genetic Results
- No results given (Active Comparator): Participants will not be offered to receive the results of genotyping for RS1051730 until all data collection has been completed.
  Interventions: Behavioral: No results given

INTERVENTIONS:
Behavioral: Receipt of Genetic Results — Participants will receive the results of genotyping for RS1051730
  Arms: Receipt of Genetic Results
Behavioral: No results given — Participants will not be offered to receive the results of genotyping for RS1051730 until all data collection has been completed.
  Arms: No results given

SUMMARY:
Innovative strategies to reduce adult smoking prevalence include using genetic information to motivate cessation and, ultimately, to tailor cessation pharmacotherapy. Success of these interventions depends, in part, on smokers' interest and participation in genetic testing related to cessation and their understanding and use of the results (i.e., their genetic literacy). The recent availability of genetic risk testing for a nicotinic acetylcholine receptor gene (CHRNA3) variant (rs105173) associated with nicotine dependence makes it highly feasible to investigate smokers' interest in and use of genetic information about nicotine dependence. Therefore, the primary purpose of this study is to determine the impact of an intervention that provides smokers with an educational session about genetic contributions to smoking and nicotine dependence plus their genotype results for rs1051730 on smoking cessation outcomes compared to those who receive only the educational session. Secondary purposes are to determine: (a) the impact of genetic education and knowing personal genotype results on genetic literacy outcomes and (b) the feasibility of recruitment and retention methods in a study addressing genotyping for nicotine dependence. Primary outcomes are cessation-related behaviors and cognitions indicating abstinence. Secondary outcomes are cognitions and emotions indicating genetic literacy. Knowledge gained from this study has the potential for clinical translation so that as genotyping becomes part of smoking cessation, health-care providers can understand and address factors influencing smokers' adaptation to genetically-informed cessation treatment. The study will use a longitudinal, repeated measures design (experimental, control; N=90; 45/group). All participants will receive a 90-minute educational session about genetic contributions for smoking and nicotine dependence and will donate a buccal swab sample for genotyping. The investigators will then randomize participants to two groups: those who receive genotyping results in a genetic counseling session (experimental) and those who do not (control). Follow-up data will be collected from both groups at baseline and weeks 2, 6, 10 after the experimental group receives genotyping results, with a brief follow-up and study termination occurring at week 12. Control group participants will be offered their genotyping results at the end of the study.

DETAILED DESCRIPTION:
The primary aim of this study is:

Aim 1. Determine the impact of knowing personal genotyping results for nicotine dependence risk on the smoking cessation (primary) outcomes at weeks 2, 6, and 10.

The working hypotheses for the cessation-related behaviors are:

1. When compared to the control group, the experimental group will have greater: (1) smoking abstinence; (2) use of formal smoking cessation programs; (3) contact with health-care provider for cessation; (4) use of pharmacotherapy, and (5) use of self-management strategies for cessation.
2. There will be no difference in the number of quit attempts between the experimental and control groups.

The working hypotheses for the cessation-related cognitions are:

1. When compared to the control group, the experimental group will have higher self-efficacy for smoking cessation.
2. When compared to the control group, the experimental group will have higher abstainer and lower smoker self-schemas.

The secondary aims are:

Aim 2. Determine the impact of knowing personal genotyping results for nicotine dependence risk on the secondary genetic literacy (secondary) outcomes at weeks 2, 6, and 10.

The working hypotheses for the genetic literacy-related cognitions and emotions are:

1. When compared to the control group, the experimental group will have greater: (1) knowledge of genetic contributions to smoking, (2) mental representations indicating endorsement of genetic risk for nicotine dependence, (3) accurate perceptions of genetic risk for nicotine dependence, and (4) self-efficacy for use of genotyping results.
2. There will be no difference in psychological distress between the experimental and control groups.

Aim 3. Explore smokers' perceptions and experiences that contextualize participation in genetic education and genotyping for nicotine dependence risk. We will conduct focus groups with both the intervention and control group participants at weeks 2 and 6 after intervention group participants receive their genotyping results.

Aim 4. Determine the feasibility of an intervention that informs people of their personal genotype results for nicotine dependence risk for a larger clinical trial, including evaluation of enrollment (recruitment efficiency, attrition, problems and solutions), intervention fidelity (delivery, receipt, enactment), data collection, subject acceptability of the intervention, and estimation of effect sizes for sample size determination in future, larger clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* >19 years of age;
* smoking>= 10 cigarettes/day;
* intention to quit smoking at some time in the future;
* able to understand, speak, and write in English, and
* physically and mentally able to participate.

The investigators are excluding participants who do not understand, speak or write in English at this time because: (1) the consent document, the educational genetics presentation, and data collection forms are currently written in English only and (2)the resources to make the educational presentation and data collection documents culturally-specific for other cultures are not available. In making the study relevant for non-English speaking participants, it is not only a literal translation the presentation and documents into another language that is needed, but the ideas of health and heredity from the culture related to the language also need to be taken into account when presenting the study and the study materials in another language.

Exclusion Criteria:

* current treatment for a mental disorder with psychotic symptoms;
* diagnosis of cancer (other than basal or squamous cell skin cancer) or other life-threatening illness;
* pregnant, or
* currently enrolled in another smoking research study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2013-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia F Houfek, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smerecnik C, Quaak M, van Schayck CP, van Schooten FJ, de Vries H. Are smokers interested in genetic testing for smoking addiction? A socio-cognitive approach. Psychol Health. 2011 Aug;26(8):1099-112. doi: 10.1080/08870446.2010.541909. Epub 2011 Jun 28. PMID 21678175
- [Background] Brock AJ, Takeda A, Brennan C, Walton RT. Treatment for tobacco dependence: a potential application for stratified medicine? Per Med. 2011 Sep;8(5):571-579. doi: 10.2217/pme.11.60. PMID 29793253
- [Background] Addicted to Nicotine: A National Research Forum. July 27-28, 1998. Bethesda, Maryland, USA. Proceedings. Nicotine Tob Res. 1999;1 Suppl 2:S1-215. No abstract available. PMID 12022131
- [Background] Fiore, M. C., Jaen, C.R., Baker, T.B., et al. (2008). Treating Tobacco Use and Dependence. 2008 Update. Clinical Practice Guideline. Rockville, MD: U.S. Department of Health and Human Services. Public Health Service.
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: current cigarette smoking among adults aged >/=18 years--United States, 2005-2010. MMWR Morb Mortal Wkly Rep. 2011 Sep 9;60(35):1207-12. PMID 21900875
- [Background] United States Department of Health and Human Services, Healthy People 2020. (2012, January 9). Tobacco Use: Objectives. Retrieved from http://healthypeople.gov/2020/topicsobjectives2020/objectiveslist.aspx?topicId=41
- [Background] Quaak M, Smerecnik C, van Schooten FJ, de Vries H, van Schayck CP. Knowledge, attitudes and preferences regarding genetic testing for smoking cessation. A cross-sectional survey among Dutch smokers. BMJ Open. 2012 Jan 5;2(1):e000321. doi: 10.1136/bmjopen-2011-000321. Print 2012. PMID 22223839
- [Background] Read CY, Perry DJ, Duffy ME. Design and psychometric evaluation of the Psychological Adaptation to Genetic Information Scale. J Nurs Scholarsh. 2005;37(3):203-8. doi: 10.1111/j.1547-5069.2005.00036.x. PMID 16235859
- [Background] Smerecnik CM, Mesters I, de Vries NK, de Vries H. Educating the general public about multifactorial genetic disease: applying a theory-based framework to understand current public knowledge. Genet Med. 2008 Apr;10(4):251-8. doi: 10.1097/GIM.0b013e31816b4ffd. PMID 18414207
- [Background] Pleasant A, McKinney J. Coming to consensus on health literacy measurement: an online discussion and consensus-gauging process. Nurs Outlook. 2011 Mar-Apr;59(2):95-106.e1. doi: 10.1016/j.outlook.2010.12.006. PMID 21402205
- [Background] Weinman J, Petrie KJ. Illness perceptions: a new paradigm for psychosomatics? J Psychosom Res. 1997 Feb;42(2):113-6. doi: 10.1016/s0022-3999(96)00294-2. No abstract available. PMID 9076639
- [Background] Brownlee, S., Leventhal, H., & Leventhal, E. A. (2000). Regulation, self-regulation, and construction of the self in maintenance of physical health. In M. Boekaerts, P.R. Pintrich, & M. Zeidner, (Eds.). Handbook of Self-Regulation. San Diego, CA: Academic Press, pp. 369-416.
- [Background] Munafo M, Clark T, Johnstone E, Murphy M, Walton R. The genetic basis for smoking behavior: a systematic review and meta-analysis. Nicotine Tob Res. 2004 Aug;6(4):583-97. doi: 10.1080/14622200410001734030. PMID 15370155
- [Background] Cervone D. The architecture of personality. Psychol Rev. 2004 Jan;111(1):183-204. doi: 10.1037/0033-295X.111.1.183. PMID 14756593
- [Background] Benowitz NL. Clinical pharmacology of nicotine: implications for understanding, preventing, and treating tobacco addiction. Clin Pharmacol Ther. 2008 Apr;83(4):531-41. doi: 10.1038/clpt.2008.3. Epub 2008 Feb 27. PMID 18305452
- [Background] Thorgeirsson TE, Geller F, Sulem P, Rafnar T, Wiste A, Magnusson KP, Manolescu A, Thorleifsson G, Stefansson H, Ingason A, Stacey SN, Bergthorsson JT, Thorlacius S, Gudmundsson J, Jonsson T, Jakobsdottir M, Saemundsdottir J, Olafsdottir O, Gudmundsson LJ, Bjornsdottir G, Kristjansson K, Skuladottir H, Isaksson HJ, Gudbjartsson T, Jones GT, Mueller T, Gottsater A, Flex A, Aben KKH, de Vegt F, Mulders PFA, Isla D, Vidal MJ, Asin L, Saez B, Murillo L, Blondal T, Kolbeinsson H, Stefansson JG, Hansdottir I, Runarsdottir V, Pola R, Lindblad B, van Rij AM, Dieplinger B, Haltmayer M, Mayordomo JI, Kiemeney LA, Matthiasson SE, Oskarsson H, Tyrfingsson T, Gudbjartsson DF, Gulcher JR, Jonsson S, Thorsteinsdottir U, Kong A, Stefansson K. A variant associated with nicotine dependence, lung cancer and peripheral arterial disease. Nature. 2008 Apr 3;452(7187):638-642. doi: 10.1038/nature06846. PMID 18385739
- [Background] Ducci F, Kaakinen M, Pouta A, Hartikainen AL, Veijola J, Isohanni M, Charoen P, Coin L, Hoggart C, Ekelund J, Peltonen L, Freimer N, Elliott P, Schumann G, Jarvelin MR. TTC12-ANKK1-DRD2 and CHRNA5-CHRNA3-CHRNB4 influence different pathways leading to smoking behavior from adolescence to mid-adulthood. Biol Psychiatry. 2011 Apr 1;69(7):650-60. doi: 10.1016/j.biopsych.2010.09.055. Epub 2010 Dec 17. PMID 21168125
- [Background] Munafo MR, Johnstone EC, Walther D, Uhl GR, Murphy MF, Aveyard P. CHRNA3 rs1051730 genotype and short-term smoking cessation. Nicotine Tob Res. 2011 Oct;13(10):982-8. doi: 10.1093/ntr/ntr106. Epub 2011 Jun 20. PMID 21690317
- [Background] Hung RJ, McKay JD, Gaborieau V, Boffetta P, Hashibe M, Zaridze D, Mukeria A, Szeszenia-Dabrowska N, Lissowska J, Rudnai P, Fabianova E, Mates D, Bencko V, Foretova L, Janout V, Chen C, Goodman G, Field JK, Liloglou T, Xinarianos G, Cassidy A, McLaughlin J, Liu G, Narod S, Krokan HE, Skorpen F, Elvestad MB, Hveem K, Vatten L, Linseisen J, Clavel-Chapelon F, Vineis P, Bueno-de-Mesquita HB, Lund E, Martinez C, Bingham S, Rasmuson T, Hainaut P, Riboli E, Ahrens W, Benhamou S, Lagiou P, Trichopoulos D, Holcatova I, Merletti F, Kjaerheim K, Agudo A, Macfarlane G, Talamini R, Simonato L, Lowry R, Conway DI, Znaor A, Healy C, Zelenika D, Boland A, Delepine M, Foglio M, Lechner D, Matsuda F, Blanche H, Gut I, Heath S, Lathrop M, Brennan P. A susceptibility locus for lung cancer maps to nicotinic acetylcholine receptor subunit genes on 15q25. Nature. 2008 Apr 3;452(7187):633-7. doi: 10.1038/nature06885. PMID 18385738
- [Background] Amos CI, Wu X, Broderick P, Gorlov IP, Gu J, Eisen T, Dong Q, Zhang Q, Gu X, Vijayakrishnan J, Sullivan K, Matakidou A, Wang Y, Mills G, Doheny K, Tsai YY, Chen WV, Shete S, Spitz MR, Houlston RS. Genome-wide association scan of tag SNPs identifies a susceptibility locus for lung cancer at 15q25.1. Nat Genet. 2008 May;40(5):616-22. doi: 10.1038/ng.109. Epub 2008 Apr 2. PMID 18385676
- [Background] Abrams, D.B., Niaura, R., Brown, R.A., Emmons, K.M., Goldstein, M.G., & Monti, P.M. (2003). The Tobacco Dependence Treatment Handbook: A Guide to Best Practices. New York: The Guilford Press.
- [Background] Quaak M, van Schayck CP, Knaapen AM, van Schooten FJ. Genetic variation as a predictor of smoking cessation success. A promising preventive and intervention tool for chronic respiratory diseases? Eur Respir J. 2009 Mar;33(3):468-80. doi: 10.1183/09031936.00056908. PMID 19251795
- [Background] Lerman CE, Schnoll RA, Munafo MR. Genetics and smoking cessation improving outcomes in smokers at risk. Am J Prev Med. 2007 Dec;33(6 Suppl):S398-405. doi: 10.1016/j.amepre.2007.09.006. PMID 18021915
- [Background] Malaiyandi V, Sellers EM, Tyndale RF. Implications of CYP2A6 genetic variation for smoking behaviors and nicotine dependence. Clin Pharmacol Ther. 2005 Mar;77(3):145-58. doi: 10.1016/j.clpt.2004.10.011. PMID 15735609
- [Background] Smerecnik C, Grispen JE, Quaak M. Effectiveness of testing for genetic susceptibility to smoking-related diseases on smoking cessation outcomes: a systematic review and meta-analysis. Tob Control. 2012 May;21(3):347-54. doi: 10.1136/tc.2011.042739. Epub 2011 Sep 26. PMID 21948804
- [Background] Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine Tob Res. 2003 Feb;5(1):13-25. PMID 12745503
- [Background] Audrain J, Boyd NR, Roth J, Main D, Caporaso NF, Lerman C. Genetic susceptibility testing in smoking-cessation treatment: one-year outcomes of a randomized trial. Addict Behav. 1997 Nov-Dec;22(6):741-51. doi: 10.1016/s0306-4603(97)00060-9. PMID 9426791
- [Background] Perkins, K.A., Conklin, C.A., & Levine, M.D. (2008). Cognitive-Behavioral Therapy for Smoking Cessation. New York: Routledge.
- [Background] Cokkinides VE, Ward E, Jemal A, Thun MJ. Under-use of smoking-cessation treatments: results from the National Health Interview Survey, 2000. Am J Prev Med. 2005 Jan;28(1):119-22. doi: 10.1016/j.amepre.2004.09.007. PMID 15626567
- [Background] Hung WT, Dunlop SM, Perez D, Cotter T. Use and perceived helpfulness of smoking cessation methods: results from a population survey of recent quitters. BMC Public Health. 2011 Jul 27;11:592. doi: 10.1186/1471-2458-11-592. PMID 21791111
- [Background] Wright AJ, Weinman J, Marteau TM. The impact of learning of a genetic predisposition to nicotine dependence: an analogue study. Tob Control. 2003 Jun;12(2):227-30. doi: 10.1136/tc.12.2.227. PMID 12773736
- [Background] Etter JF, Bergman MM, Humair JP, Perneger TV. Development and validation of a scale measuring self-efficacy of current and former smokers. Addiction. 2000 Jun;95(6):901-13. doi: 10.1046/j.1360-0443.2000.9569017.x. PMID 10946439
- [Background] Liang, K.Y, & Zeger, S.L. (1986). Longitudinal data analysis using generalized linear models. Biometrika, 73, 13-22
- [Background] Weinman, J., Petrie, K.J., Moss-Morris, R., & Horne, R. (1996). The illness perception questionnaire: A new method for assessing cognitive representations of illness. Psychology & Health, 11, 431-445.
- [Background] Velicer WF, Diclemente CC, Rossi JS, Prochaska JO. Relapse situations and self-efficacy: an integrative model. Addict Behav. 1990;15(3):271-83. doi: 10.1016/0306-4603(90)90070-e. PMID 2378287
- [Background] SRNT Subcommittee on Biochemical Verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002 May;4(2):149-59. doi: 10.1080/14622200210123581. No abstract available. PMID 12028847
- [Background] Doak LG, Doak CC, Meade CD. Strategies to improve cancer education materials. Oncol Nurs Forum. 1996 Sep;23(8):1305-12. PMID 8883075
- [Background] McBride CM, Bepler G, Lipkus IM, Lyna P, Samsa G, Albright J, Datta S, Rimer BK. Incorporating genetic susceptibility feedback into a smoking cessation program for African-American smokers with low income. Cancer Epidemiol Biomarkers Prev. 2002 Jun;11(6):521-8. PMID 12050092
- [Background] Cohen, J. (1988). Statistical Power Analysis for the Behavioral Sciences. Mahwah, NJ: Lawrence Erlbaum Associates, Inc.
- [Background] Lerman C, Gold K, Audrain J, Lin TH, Boyd NR, Orleans CT, Wilfond B, Louben G, Caporaso N. Incorporating biomarkers of exposure and genetic susceptibility into smoking cessation treatment: effects on smoking-related cognitions, emotions, and behavior change. Health Psychol. 1997 Jan;16(1):87-99. doi: 10.1037//0278-6133.16.1.87. PMID 9028818
- [Background] Spielberger, C.D. (1995b). Preliminary Manual for the State-Trait Personality Inventory (STPI). Unpublished manual.
- [Background] Spielberger, C.D. (1995a). Scoring information for the revised STPI. Tampa: Center for Research in Behavioral Medicine and Health Psychology, University of South Florida.
- [Background] Wright AJ, French DP, Weinman J, Marteau TM. Can genetic risk information enhance motivation for smoking cessation? An analogue study. Health Psychol. 2006 Nov;25(6):740-52. doi: 10.1037/0278-6133.25.6.740. PMID 17100502
- [Background] Sanderson SC, Michie S. Genetic testing for heart disease susceptibility: potential impact on motivation to quit smoking. Clin Genet. 2007 Jun;71(6):501-10. doi: 10.1111/j.1399-0004.2007.00810.x. PMID 17539899
- [Background] Cameron LD, Marteau TM, Brown PM, Klein WM, Sherman KA. Communication strategies for enhancing understanding of the behavioral implications of genetic and biomarker tests for disease risk: the role of coherence. J Behav Med. 2012 Jun;35(3):286-98. doi: 10.1007/s10865-011-9361-5. Epub 2011 Jun 23. PMID 21698440
- [Background] Sanderson SC, Waller J, Humphries SE, Wardle J. Public awareness of genetic influence on chronic disease risk: are genetic and lifestyle causal beliefs compatible? Public Health Genomics. 2011;14(4-5):290-7. doi: 10.1159/000294280. Epub 2010 Apr 29. PMID 20431275
- [Background] Henderson BJ, Maguire BT. Three lay mental models of disease inheritance. Soc Sci Med. 2000 Jan;50(2):293-301. doi: 10.1016/s0277-9536(99)00286-5. PMID 10619697
- [Background] Moss-Morris, R., Weinman, J., Petrie, K.J., Horne, R., Cameron, L.D., & Buick, D. (2002). The revised illness perception questionnaire (IPQ-R). Psychology & Health, 17, 1-16.
- [Background] Condit CM. Public understandings of genetics and health. Clin Genet. 2010 Jan;77(1):1-9. doi: 10.1111/j.1399-0004.2009.01316.x. PMID 20092586
- [Background] Smerecnik CM, Mesters I, de Vries NK, de Vries H. Applying a theory-based framework to understand public knowledge of genetic risk factors: a case for the distinction between how-to knowledge and principles knowledge. Public Health Genomics. 2011;14(4-5):259-70. doi: 10.1159/000294149. Epub 2010 Mar 12. PMID 20224242
- [Background] Park ER, Kleimann S, Youatt EJ, Lockhart A, Campbell EG, Levy DE, Halbert CH, Schmieder E, Krishna R, Shields AE. Black and White adults' perspectives on the genetics of nicotine addiction susceptibility. Addict Behav. 2011 Jul;36(7):769-72. doi: 10.1016/j.addbeh.2011.02.007. Epub 2011 Feb 25. PMID 21406316
- [Background] Shadel WG, Mermelstein R, Borrelli B. Self-concept changes over time in cognitive-behavioral treatment for smoking cessation. Addict Behav. 1996 Sep-Oct;21(5):659-63. doi: 10.1016/0306-4603(95)00088-7. PMID 8876764
- [Background] Cappella, J.N., Lerman, C., Romantan, A., & Baruh, L. (2003). News about genetics and smoking. Communications Research, 32, 478-502.
- [Background] Hendricks PS, Delucchi KL, Hall SM. Mechanisms of change in extended cognitive behavioral treatment for tobacco dependence. Drug Alcohol Depend. 2010 Jun 1;109(1-3):114-9. doi: 10.1016/j.drugalcdep.2009.12.021. Epub 2010 Jan 21. PMID 20096510

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 169 persons contacted the study coordinator (n = 169). Of these, 63 were lost to follow-up due to non-return of phone call when contacted. A total of 43 participants completed the assessment for eligibility. Of these 19 were excluded (7 did not meet the criteria and 12 declined to participate further). A total of 24 participants were randomized, 12 each to the experimental and control groups.
Period: Overall Study
Arm/Group | Receipt of Genetic Results | No Results Given
Started | 12 | 12
Completed | 8 (Nine participants obtained genotyping results. Eight participants provided follow-up data.) | 11 (Six participants received genotyping results that were offered upon study completion. Eleven participants provided follow-up data.)
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Receipt of Genetic Results | No Results Given | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 11 | 9 | 20
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Participant Demographic Data
  Participants
    United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Smoking Abstinence at 6 and 10 Weeks After Genotyping Results
Description: Abstinence: Point-Prevalence & Continuous Self-Report; Exhaled Carbon Monoxide (CO): <= 6 ppm past 24 hrs.; Salivary Cotinine: <15 ng/ml past 7 days
Time Frame: Assessed at Weeks 6 and 10 after Genotyping Results, Week 10 reported
Measure: Count of Participants; unit: Participants
Arm/Group | Receipt of Genetic Results | No Results Given
Number analyzed (Participants) | 8 | 11
Participants
  Total Achieving Cessation | 1 | 0
  Total Still Smoking | 7 | 11

2. Secondary Outcome: Change in Baseline Use of Pharmacotherapy at 6 and 10 Weeks After Genotyping Results
Description: Use of Pharmacotherapy: Self-report of type and frequency of use of FDA-approved smoking cessation medications.
Time Frame: Assessed at Weeks 6 and 10 weeks after Genotyping Results, Week 10 reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Receipt of Genetic Results | No Results Given
Number analyzed (Participants) | 8 | 11
Participants
  Pharmacotherapy use | 2 | 2
  No pharmacotherapy use | 6 | 9
Statistical Analysis 1: Comparison: Receipt of Genetic Results vs No Results Given; Test type: Other; Frequencies and percentages were used to determine this secondary outcome

ADVERSE EVENTS:
Time Frame: Baseline through follow-up (10 weeks)
Arm/Group | Receipt of Genetic Results | No Results Given
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Recruitment goals were not met. Only 14% of those who inquired about the study enrolled. Most individuals who did not participate were interested in a smoking cessation study and/or a higher honorarium. Data collection times were streamlined to encourage continued study participation, which was successful. Recommendations include: (1) offering a smoking cessation component and (2) better explaining the practical benefit of knowing genetic risk for nicotine dependence during recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No